CLINICAL TRIAL: NCT02576912
Title: Testing the Interactive Effects of Delta-9-Tetrahydrocannabinol and Pregnenolone
Acronym: THC-Preg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1501015242
Record Dates: First submitted 2015-03-24; First posted 2015-10-15 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Cannabis; Marijuana; THC; Pregnenolone; Psychotic Disorders; PREG
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active Delta-9-THC and Placebo Pregnenolone (Experimental)
  Interventions: Drug: Active Delta-9-THC; Drug: Placebo
- Active Delta-9-THC and Active Pregnenolone (Experimental)
  Interventions: Drug: Active Delta-9-THC; Drug: Active Pregnenolone
- Placebo Delta-9-THC and Active Pregnenolone (Experimental)
  Interventions: Drug: Active Pregnenolone; Drug: Placebo
- Placebo Delta-9-THC and Placebo Pregnenolone (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active Delta-9-THC — Active Delta-9-THC (0.036 mg/kg) given intravenously.
  Arms: Active Delta-9-THC and Active Pregnenolone; Active Delta-9-THC and Placebo Pregnenolone
Drug: Active Pregnenolone — A dose given sublingually.
  Arms: Active Delta-9-THC and Active Pregnenolone; Placebo Delta-9-THC and Active Pregnenolone
Drug: Placebo — A placebo dose given sublingually.
  Arms: Active Delta-9-THC and Placebo Pregnenolone; Placebo Delta-9-THC and Placebo Pregnenolone
Drug: Placebo — Placebo dose given intravenously.
  Arms: Placebo Delta-9-THC and Active Pregnenolone; Placebo Delta-9-THC and Placebo Pregnenolone

SUMMARY:
The overall purpose of this study is to examine the effect of pregnenolone (PREG) on the acute psychosis-like and cognitive effects of Delta-9-tetrahydrocannabinol (THC). This will be tested by pretreating healthy individuals with PREG and then assessing their responses to THC.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to cannabis at least once in lifetime.

Exclusion Criteria:

* Cannabis naive
* Individuals with a documented reaction/allergy to Pregnenolone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02; Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Baseline, +110, +180, and +240 minutes after start of THC Infusion
  Positive, negative, and general symptoms will be assessed using the positive, negative, and general symptom subscales of the PANSS.

SECONDARY OUTCOMES:
Clinician Administered Dissociative Symptoms Scale (CADSS) | Baseline; +15, +110, +180, and +240 minutes after start of THC infusion
  Perceptual alterations will be measured using the CADSS. This is a scale consisting of 19 self-reported items and 9 clinician-rated items. The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.
Visual Analog Scale (VAS) | Baseline; +15, +110, +180, and +240 minutes after start of THC infusion
  Feeling states associated with cannabis intoxication will be measured using a self-reported visual analog scale of feeling states associated with cannabis effects (ex: "high," "calm," "anxious"). Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 11mm line. These data will be captured to validate that the experiment is relevant to cannabis effects.
Psychotomimetic States Inventory (PSI) | Baseline; +110, +180, and +240 minutes after start of THC infusion
  The PSI is a measure of drug induced psychotomimetic states. This self-reported scale consists of 28 items rated 0 (not at all) to 3 (extremely) and will facilitate the characterization of a wide range of dissociative/hallucinatory phenomena as well as cognitive disorganization associated with the administration of THC.
Cognitive Test Battery | 25 minutes after start of THC infusion
  Several computer tasks will be administered in order to evaluate the effects of cannabis on verbal learning and memory, visual recognition, spatial working memory, and working memory. The battery consists of five computer tasks that lasts no longer than 20 minutes in total.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD, Principal Investigator — Yale University
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States